CLINICAL TRIAL: NCT06250322
Title: A Multicenter, Observational, Single Arm Study of the TECNIS Presbyopia-correcting Intraocular Lens
Status: Completed | Type: Observational
Sponsor: Johnson & Johnson Surgical Vision, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PCOL204APME
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Cataracts
MeSH Terms: conditions — Cataract | interventions — Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Intervention — No study treatments will be administered during this study. However, data will be collected from medical records of patients who have been treated with the subject device of this study.

SUMMARY:
Ambispective post-market data collection on visual symptoms, patient satisfaction and surgeon experience with the TECNIS PC IOL.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are bilaterally implanted with TECNIS PC IOL and are at least 45 days postoperative from their second eye surgery
* Clear intraocular media
* Signed informed consent and data protection documentation
* Availability, willingness, ability, and sufficient cognitive awareness to comply with examination procedures
* Ability to understand, read, and write English or the local language in which the informed consent and questionnaires are provided

Exclusion Criteria:

* Subjects with ongoing adverse events that might impact outcomes during the study
* Use of systemic or ocular medication that may affect vision
* Acute or chronic disease or condition, ocular trauma or surgery that may confound results
* Patients with amblyopia, strabismus, nystagmus
* Concurrent participation in another clinical trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A pre-existing population of subjects bilaterally implanted with the PC IOL at approximately 20 sites in Europe and Asia Pacific. Bilateral pseudophakic subjects implanted with the TECNIS PC IOL will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 307 (Actual)
Dates: Start 2024-04-10 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Visual Symptoms | 3month postoperative
  Patient questionnaires
Surgeon Experience | 3month postoperative
  Questionnaire
Visual Acuity | 3month postoperative
  Visual Acuity will be collected with standard clinical charts.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Surgical Vision, Inc. Clinical Trial, Study Director — Johnson & Johnson Surgical Vision, Inc.
Locations (20):
- Australia (4):
  - Vision Eye Institute, Chatswood, New South Wales
  - Sunshine Eye Clinic, Birtinya, Queensland
  - The Queensland Eye Institute Foundation, Woolloongabba, Queensland
  - Lions Eye Institute, Nedlands, Western Australia
- Vienna Institute for Research in Ocular Surgery - A Karl-Landsteiner-Institute, Vienna, Austria
- France (2):
  - CHU Morvan Brest, Brest
  - Clinique Juge Marseille, Marseille
- Germany (2):
  - Augenklinik Ahaus GmbH & Co. KG, Ahaus
  - Augenklinik Dardenne, Bonn
- India (4):
  - Narayana Nethralaya, Bengaluru
  - The Eye Foundation, Coimbatore
  - Centre for Sight Eye Institute, New Delhi
  - All India Institute of Medical Sciences (AIIMS), New Delhi
- Netherlands (2):
  - Oogziekenhuis Rotterdam, Rotterdam
  - ETZ, Tilburg
- South Korea (2):
  - Kim's eye clinic, Seoul
  - Korea Uni.Kuro, Seoul
- Spain (3):
  - Clinica Oftalmologica Diez del Corral, Madrid
  - Mirzana IOA, Madrid
  - Vithas Alicante, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu